CLINICAL TRIAL: NCT02873078
Title: Internet-Delivered Cognitive Behavior Therapy for Children With Functional Abdominal Pain Disorders - a Randomized Controlled Trial
Brief Title: Internet-Delivered CBT for Children With Functional Abdominal Pain Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ola Olen, MD PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT ICBT FAPD
Record Dates: First submitted 2016-08-09; First posted 2016-08-19 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Functional Abdominal Pain Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-delivered CBT (Experimental): Children and parents will receive 10 weekly modules of cognitive behavior therapy (CBT). Parents will also receive 10 weekly modules. Main components in the children's modules are exposure for abdominal symptoms, feared stimuli and situations in which the children are afraid of having symptoms. The parental receive information on how they can support their children in the treatment and how to reinforce health y behaviors and decrease attention to pain behaviors. Therapist support is provided through written messages within the secure platform.
  Interventions: Behavioral: Internet-delivered Cognitive behavior therapy
- Waiting list (No Intervention): This is a wait-list control where the children and parents are allowed to carry on with any contacts within the health-care system, exempt for psychological treatments.

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive behavior therapy — The treatment is delivered via an online platform and is based on interventions for adults, adolescents and children tested in previous trials. Therapists are CBT-psychologists och students in clinical psychology under supervision.
  Arms: Internet-delivered CBT

SUMMARY:
This randomized controlled study aims to evaluate the efficacy of exposure-based Internet-delivered cognitive behavior therapy for children 8-12 years with Functional Abdominal Pain Disorders. The children participate along with their parents, who will also receive specific modules with information on how to support their children in the treatment. Predictors and mediators for treatment effects will be studied as well as the cost effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-12 years with either irritable bowel syndrome, functional dyspepsia or functional abdominal pain - not otherwise specified diagnosed according to Rome-III or Rome-IV criteria.
* Psychopharmacological medication stable for at least a month if medicating.
* Child and at least one parent speaking and writing swedish.
* Access to computer with Internet connection.

Exclusion Criteria:

* Severe somatic disorder and/or if the child fulfills criteria of other disorder that better explains the abdominal symptoms.
* Severe psychiatric or social problems that needs other care.
* Ongoing psychological treatment.
* School absenteeism more than 40 %.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-08; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
PedsQL Gastro | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.

SECONDARY OUTCOMES:
Faces Pain Rating Scale | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in pain intensity measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Faces Pain Rating Scale | Weekly during treatment (treatment week 1-9).
  Change in pain intensity measured with a self-rating scale weekly during treatment for mediation analyses.
Faces Pain Rating Scale rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's pain intensity measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Faces Pain Rating Scale rated by parents | Weekly during treatment (treatment week 1-9).
  Change in pain intensity measured with a self-rating scale weekly during treatment for mediation analyses.
PedsQL Gastro rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child gastrointestinal symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
PedsQL Gastro rated by parents | Weekly during treatment (treatment week 1-9).
  Change in child gastrointestinal symptoms measured with a self-rating scale weekly during treatment for mediation.
Pediatric quality of life inventory (PedsQL QOL) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in quality of life measured measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Pediatric quality of life inventory (PedsQL QOL) rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child quality of life measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Painfree days | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in pain free days measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Painfree days | Weekly during treatment (treatment week 1-9)
  Change in pain free days measured with a self-rating scale weekly during treatment for mediation analyses.
Painfree days rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's pain free days measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Painfree days rated by parents | Weekly during treatment (treatment week 1-9)
  Change in child's pain free days measured with a self-rating scale weekly during treatment for mediation analyses.
IBS-Behavioral responses questionnaire (IBS-BRQ) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in childs behavioral responses to abdominal symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
IBS-Behavioral responses questionnaire (IBS-BRQ) | Weekly during treatment (treatment week 1-9)
  Change in child's behavioral responses to abdominal symptoms measured with a self-rating scale weekly during treatment for mediation analyses.
IBS-Behavioral responses questionnaire (IBS-BRQ) parental version | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's behavioral responses to abdominal symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
IBS-Behavioral responses questionnaire (IBS-BRQ) parental version | Weekly during treatment (treatment week 1-9)
  Change in child's behavioral responses to abdominal symptoms measured with a self-rating scale weekly during treatment for mediation analyses.
Spence Children Anxiety Scale - short version (SCAS-S) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's anxiety symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Spence Children Anxiety Scale - short version (SCAS-S) rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's anxiety symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Child Depression Inventory - short version (CDI-S) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's depressive symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Visceral Sensitivity Index | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in visceral sensitivity measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Visceral Sensitivity Index | Weekly during treatment (treatment week 1-9)
  Change in visceral sensitivity measured with a self-rating scale weekly during treatment for mediation analyses.
Client Satisfactory Questionnaire (CSQ) | At week 10
  Client satisfaction rated measured with a self-rating scale
Client Satisfactory Questionnaire (CSQ) rated by parents | At week 10
  Client satisfaction rated measured with a self-rating scale
Subjective Assessment Questionnaire (SAQ) | At week 10
  Subjective change in symptoms measured with a self-rating scale
Subjective Assessment Questionnaire (SAQ) rated by parents | At week 10
  Subjective change in the child's symptoms measured with a self-rating scale by the parents.
Rome-IV questionnaire | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in diagnostic status of functional abdominal pain disorder measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Kidscreen | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in quality of life for use in economic evaluation measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
School absenteeism rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's school absenteeism measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
School absenteeism rated by parents | Weekly during treatment (treatment week 1-9)
  Change in child's school absenteeism measured with a self-rating scale weekly during treatment for mediation analyses.
Pain Catastrophizing Scale, parental version (PCS-P) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in parental catastrophizing of the child's symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Pain Catastrophizing Scale, parental version (PCS-P) | Weekly during treatment (treatment week 1-9)
  Change in parental catastrophizing of the child's symptoms measured with a self-rating scale weekly during treatment for mediation analyses.
Children´s Somatization Inventory (CSI 24) rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in child's somatization symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Adverse events (AE) | At week 10
  Adverse events during treatment measured with a self-rating scale by the parents.
Working Alliance Inventory (WAI) short version | At week 4
  Working alliance in first three weeks of treatment measured with a self-rating scale by the parents.
The treatment credibility scale rated by parents. | At week 2
  Treatment credibility measured with a self-rating scale by the parents.
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) rated by parents | Baseline, at weeks 3, 7, 10 and at 9 months
  Costs associated with the disorder measured with a self-rating scale by the parents.
General health questionnaire (GHQ-12) rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in general health measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Generalised anxiety disorder assessment (GAD 7) rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in parental anxiety symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Adult responses to children's symptoms (ARCS) rated by parents | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months
  Change in parental responses to child's symptoms measured with a self-rating scale from baseline to 10 weeks, from baseline to 9 months, and from baseline to 15 months for analysis of effect.
Adult responses to children's symptoms (ARCS) rated by parents | Weekly during treatment (treatment week 1-9)
  Change in parental responses to child's symptoms measured with a self-rating scale weekly during treatment for mediation analyses.
PedsQL Gastro | Weekly during treatment (treatment week 1-9).
  Change in gastrointestinal symptoms measured with a self-rating scale weekly during treatment for mediation analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Olén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Child and Adolescent Psychiatry in Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lalouni M, Ljotsson B, Bonnert M, Ssegonja R, Benninga M, Bjureberg J, Hogstrom J, Sahlin H, Simren M, Feldman I, Hedman-Lagerlof E, Serlachius E, Olen O. Clinical and Cost Effectiveness of Online Cognitive Behavioral Therapy in Children With Functional Abdominal Pain Disorders. Clin Gastroenterol Hepatol. 2019 Oct;17(11):2236-2244.e11. doi: 10.1016/j.cgh.2018.11.043. Epub 2018 Nov 28. PMID 30502501